CLINICAL TRIAL: NCT06765421
Title: Optimising General Practice Long COVID Care - Feasibility Trial of a Pilot Educational Intervention.
Brief Title: Optimising General Practice Long COVID Care - an Educational Intervention.
Acronym: GP-COV-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: HRB Primary Care Clinical Trials Network Ireland (Unknown); Mater Misericordiae University Hospital (Other); Irish College of General Practitioners (Unknown); St Vincent's University Hospital, Ireland (Other); Health Services Executive, Ireland (Unknown); South East Technological University, Ireland (Unknown); National Rehabilitation Hospital, Dublin, Ireland (NRH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R27255
Record Dates: First submitted 2024-12-12; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Long COVID
Keywords: Feasibility Studies; General Practice; long COVID; Pilot Study; Medical Education
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): GP practices in the intervention group will be provided with a 'long COVID Toolkit for GPs', they will be invited to attend an long COVID educational webinar, and they will be asked to perform a detailed case review of patients enrolled in the study.
  Interventions: Behavioral: Intervention Group
- Control group (No Intervention): Control group GPs will be asked to deliver care as usual for patients enrolled in the study.

INTERVENTIONS:
Behavioral: Intervention Group — Intervention group activity involves three components:
  1. Intervention group GPs will be provided with a long COVID 'toolkit'. The toolkit will be prepared by the study team in collaboration with expert clinicians and public and patient representatives as a resource for GPs to use in patient care.
  2. GPs will attend an expert clinician / patient led long COVID educational session grounded in the findings of the toolkit.
  3. Applying learnings to date, each GP will conduct case reviews of eight patients with long COVID attending their practice and provide patient care as appropriate.
  Arms: Intervention group

SUMMARY:
This trial will evaluate the feasibility of a pilot educational intervention for GPs that aims to enhance care and care outcomes among patients with long COVID at six general practices in the Ireland East region.

Our first objective is to conduct focus groups with key stakeholders (GPs, other health professionals, patients, families/carers) that will inform the contents of an education intervention. The second objective will be to implement this educational intervention, and the third objective will be to determine whether the intervention is feasible.

Study outcomes will include:

* Qualitative findings from co-design focus groups and post-intervention semi-structured interviews with GPs.
* Practice and patient study recruitment and retention data.
* GP / Practice characteristics: age & gender, practice location, general and COVID-19 patient population figures.
* Patient characteristics: Patient age, gender, COVID-19 vaccination status, and medical history details.
* Patient scores on a self-report measure assessing the symptoms, symptom severity, functional impact, and overall health (COVID-19 Yorkshire Rehabilitation Scale (C-19-YRS)).

ELIGIBILITY:
Inclusion Criteria:

1. Age: Aged 18 years or older at the time of enrolment.
2. Registration: Are registered as patients at the study's participating practices.
3. COVID-19 Diagnosis:

   * Previously received a positive COVID-19 PCR or antigen test, or
   * Previously been clinically diagnosed with COVID-19 by a healthcare provider.
4. Persistent Symptoms:

   o Have spoken with their general practitioner (GP) about experiencing persistent symptoms lasting four weeks or more since their COVID-19 diagnosis.
5. Consent: Willing and able to provide informed consent to participate in the study.

Exclusion Criteria:

1. Vulnerability: Deemed by participating GPs to be a vulnerable individual whose best interests are served by not participating in the study, such as (but not limited to):

* People with language difficulties that prevent meaningful communication.
* Individuals with a recognised or diagnosed intellectual, physical, or mental impairment.
* Older adults considered particularly vulnerable.
* Individuals residing in institutions (e.g., care homes or prisons).
* Individuals with an unequal relationship with the researcher(s) (e.g., hierarchical dependence).
* Members of marginalised or disadvantaged groups for whom participation may present undue burden or risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Qualitative data from focus groups and post-intervention interviews | Focus groups (4 weeks), post intervention interviews (4 weeks).
  Qualitative analyses will be used to capture focus group and intervention participants' study related views and experiences, with emphasis on accounts illustrating the intervention's feasibility.

SECONDARY OUTCOMES:
Study engagement data | 12 weeks
  Descriptive statistics will assess trends relating to study invitation, commencement, and completion. Qualitative analysis will examine reasons for study exclusion, non-commencement, and non-completion.
GP and patient demographics / medical details | 4 weeks
  Descriptive statistics and qualitative analysis of open-ended responses outlining practice, GP, and patient demographics, as well as patient medical details, will be conducted.
Patients'scores on the COVID-19-YRS | 6 weeks
  Descriptive and inferential statistics outlining aggregated baseline and six-week follow-up scores on the The Covid-19 Yorkshire Rehabilitation Scale (C-19-YRS) will be calculated. The C19-YRS has four subscales concerned with the severity of patients' key symptoms, functional limitations, overall health, and additional symptoms. Each item is rated on a 0-10 numerical rating scale, where 0 represents the symptom not being present, and 10 represents the symptom being extremely severe or life disturbing.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Cullen, MD, Principal Investigator — UCD NUI: University College Dublin

IPD SHARING:
Plan to Share IPD: Undecided